CLINICAL TRIAL: NCT07300085
Title: A Phase 1, Double-blind, Randomized Trial to Evaluate Safety and Immunogenicity of Fluzone® High-Dose Influenza Vaccine When Concomitantly Administered With CD388, a Novel Long-Acting Antiviral Conjugate for the Prevention of Influenza
Brief Title: A Trial to Evaluate the Effect of CD388 on the Immunogenicity of Fluzone® HD Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD388.SQ.1.08
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Influenza; Antiviral Agents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluzone HD plus CD388 (Experimental): Participants will be randomized to receive open-label Fluzone HD influenza vaccine by intramuscular (IM) injection plus CD388 450 milligrams (mg) by subcutaneous (SQ) injection. Participants will be randomized at a 1:1 ratio between the 2 arms.
  Interventions: Biological: Fluzone HD influenza vaccine; Combination Product: CD388 Injection
- Fluzone HD plus Placebo (Placebo Comparator): Participants will be randomized to receive open-label Fluzone HD influenza vaccine by IM injection plus placebo by SQ injection. Participants will be randomized at a 1:1 ratio between the 2 arms.
  Interventions: Biological: Fluzone HD influenza vaccine; Combination Product: Placebo

INTERVENTIONS:
Biological: Fluzone HD influenza vaccine — Fluzone HD injectable suspension, 2025-2026 Formula
Combination Product: CD388 Injection — CD388 liquid for injection
  Arms: Fluzone HD plus CD388
Combination Product: Placebo — Placebo to match
  Arms: Fluzone HD plus Placebo

SUMMARY:
The goal of this clinical study is to investigate how safe and effective it is to receive both the Fluzone® High-Dose (HD) influenza vaccine and CD388, a long-acting antiviral medicine, at the same time. Some participants will receive the vaccine and CD388, while others will receive the vaccine and a placebo. The study aims to determine whether taking CD388 together with the flu vaccine affects the body's ability to build protection-called an immune response-against the flu, as compared to getting the vaccine with a placebo. The hypothesis is that giving both at the same time does not weaken the immune response to the vaccine. The study will measure the amount of antibodies (proteins produced by the immune system to fight flu viruses) generated by participants in both groups to check that CD388 does not interfere with how well the vaccine works. Participants will also be closely watched for any side effects or reactions to check that CD388 is safe to take alongside the vaccine. Expanded access to the study treatments (flu vaccine and CD388) will not be provided to participants after the study ends.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized trial to evaluate the immunogenicity of Fluzone® HD influenza vaccine when concomitantly administered with either CD388 or placebo, in healthy participants. This study will also evaluate the safety and tolerability of CD388 when administered with Fluzone HD compared to Fluzone HD with placebo. The pharmacokinetics (PK) of CD388 in plasma when administered concomitantly with Fluzone HD vaccine will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 to ≤ 49 years of age at the time of signing the informed consent.
2. Be able to understand and comply with the trial procedures, understand the risks involved in the trial, and provide written informed consent before the first trial-specific procedure.
3. Be deemed healthy by the Investigator, as determined via medical history and clinical examination before enrolling in the trial.
4. Be able to complete all screening period evaluations and attend the required follow-up visits at the site.
5. Have not received any seasonal influenza vaccine and have not had a diagnosed or suspected influenza infection within 12 months prior to Day 1 of the trial, based on participant self-report.
6. Have a body mass index (BMI; calculated as weight in kilograms [kg] divided by height in meters [m] squared)) between 18 and 32 kg/m^2, inclusive, and body weight not less than 50 kg at screening.
7. Have resting vital signs at screening within the following ranges:

   1. Systolic blood pressure ≥100 millimeters of mercury (mmHg)
   2. Diastolic blood pressure ≥50 mmHg
   3. Heart rate (HR) ≤100 beats per minute Note: If vital signs are outside of the above ranges, the Investigator may obtain up to two additional readings within the screening period.
8. Have a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at screening, including: HR between 45 and 100 bpm (inclusive); QT interval corrected using Fridericia's formula (QTcF) ≤ 450 milliseconds (ms) for males and ≤ 470 ms for females; QRS interval <120 ms; PR interval <220 ms; and morphology consistent with healthy cardiac conduction.
9. Be a nonsmoker within the previous 6 months before screening, and does not use tobacco-containing, or nicotine-containing products, including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, e-cigarettes, nicotine patch, or nicotine gum.
10. Have a negative urine drug screen for drugs of abuse at screening and on Pre-Dose Day 1. The presence of marijuana or tetrahydrocannabinol (THC) in the urine is not exclusionary unless the Investigator determines that the participant's marijuana or THC use qualifies as substance abuse.
11. Be willing to abstain from alcohol, recreational drugs, and tobacco-containing and nicotine-containing products throughout their participation in the trial.
12. Have clinical chemistry, hematology, and complete urinalysis results at screening within the reference range for the testing laboratory unless the out-of-range results are deemed not clinically significant by the Investigator.
13. Be seronegative for hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (HCV Ab), and human immunodeficiency virus (HIV) antibody at screening.
14. Must agree to the following contraception requirements:

    a. Females of childbearing potential must use a highly effective, preferably user-independent, method of contraception (failure rate of less than 1 percent per year when used consistently and correctly) from ≥2 weeks prior to enrollment and agree to remain on a highly effective method from Day 1 until 40 weeks after trial intervention administration. Note: A female is considered of childbearing potential (i.e., fertile) following menarche and until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in females not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

    Note: Contraceptive (birth control) use by participants should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.
15. Must agree not to donate blood from Day 1 until 40 weeks after administration of trial intervention.
16. Must be able to read, understand, and complete trial questionnaires and diary entries (paper or electronic), and, if the electronic format is used, be able to work with smartphones, tablets, or computers as applicable. Must also be willing and able to adhere to the prohibitions and restrictions specified in the protocol. If no appropriate language version of the diary or questionnaires (paper or electronic) is available, the participant should not be enrolled.
17. Must be willing to provide verifiable identification, has means to be contacted, and is able to contact the Investigator/trial site and communicate reliably during participation in this trial.

Exclusion Criteria:

1. Has a condition that the Investigator believes would interfere with the participant's ability to provide written informed consent, comply with trial instructions, or which might confound the interpretation of the trial results or put the participant at undue risk.
2. Have a current or past history of a clinically significant cardiovascular, cerebrovascular, respiratory, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the Investigator.
3. Had an active malignancy within 5 years prior to screening, except basal cell or squamous cell skin cancer. Any history of breast cancer or melanoma is exclusionary.
4. Have a history of any drug abuse within 1 year prior to screening or has used any hard drugs (such as cocaine, phencyclidine [PCP], natural and synthetic opiates, and amphetamine derivatives) within 1 year prior to screening. Individuals that have taken an opioid or amphetamine medication within the previous year prior to screening that was prescribed by a healthcare provider will not be excluded unless they are currently taking the medication at the time of screening.
5. Have a history of regular alcohol consumption exceeding 14 drinks/week (1 drink equals 5 ounces [150 milliliters {mL}] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening or alcohol abuse within 1 year prior to screening.
6. Are taking or have received any of the following:

   1. Medications, Supplements, Herbals (within 14 days): Any prescription or over-the-counter medication, vitamin, dietary supplement, or herbal product with known or suspected immunomodulatory effects within 14 days prior to Day 1, unless approved in advance by the Principal Investigator or sponsor medical monitor. The use of chronic, stable medications for non-immunomodulating indications (e.g., antihypertensive agents, thyroid replacement, oral contraceptives) is permitted if the regimen has been stable for at least 30 days prior to Day 1, with medical monitor approval. Any medication prescribed should be cross-referenced to ensure it is not prescribed for an exclusionary condition.
   2. Vaccinations (within 14 days): Any vaccination within 14 days prior to Day 1. Receipt of any influenza vaccine within 12 months prior to Day 1 is exclusionary. Note: Vaccines include, but are not limited to, COVID-19, pneumococcal, varicella, meningococcal, rubella, measles, mumps, hepatitis B, tetanus, and other routine or investigational vaccines.
   3. Immune Serum Globulin (6 weeks): Has received any immune serum globulin or blood-derived products within 6 weeks prior to Day 1.
   4. Immunosuppressive/Immunomodulatory Therapy (6 weeks): Any systemic corticosteroid therapy (oral or parenteral, equivalent to ≥10 mg/day prednisone for more than 14 consecutive days) or any other immunosuppressive or immunomodulatory agent within 6 weeks prior to Day 1. NOTE: Topical, inhaled, or intranasal corticosteroids at low- to moderate-dose regimens are permitted if not intended for immune suppression and at stable doses for ≥30 days before Day 1.
7. Have a contraindication to Fluzone HD or CD388 or any of the excipients and/or history of a clinically significant allergic or anaphylactic reaction to any medication or following influenza vaccination.
8. Has previously been diagnosed with Guillain-Barre Syndrome following a previous influenza vaccination.
9. Have previously participated in a clinical trial in which CD388 was a trial intervention.
10. Has participated in other trials involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before screening for the current trial and during participation in the current trial.
11. Has a positive rapid antigen test result for either Coronavirus disease 2019 (COVID-19)/severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or for influenza at Pre-Dose Day 1.
12. Has donated ≥450 mL of blood (1 unit) within 2 months before entering the trial or planning to donate blood during the trial or within 36 weeks after the final visit.
13. Have a known or suspected allergy or history of anaphylaxis to zanamivir (following administration of inhaled or intravenous formulations), monoclonal antibodies (including Fc domains), or any of the components of CD388.
14. Had major surgery (e.g., cardiac, pulmonary, neurologic, or abdominal operations) within 4 weeks prior to screening, or will not have fully recovered from such prior surgery; or has major surgery planned during the time the participant is expected to participate in this trial.
15. Have any finding (at the time of screening) that may significantly increase the risk of participation in this trial, affect the ability to participate in this trial, or impair interpretation of the trial data.
16. Have current or planned participation in another clinical trial where trial intervention is being administered while participating in this current trial.
17. Have a contraindication to SQ or IM injections and venipunctures (e.g., bleeding disorders).
18. Are currently pregnant or breastfeeding, intends to become pregnant or breastfeed, or has a positive pregnancy test during the screening period.
19. Has direct involvement in this proposed trial or other studies under the direction of the Investigator, sub-investigators, or trial site personnel; is a family member of an individual with such direct involvement; or is an employee of the Sponsor.
20. In the opinion of the Investigator, is unlikely to adhere to the requirements of this trial.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Immune Responses in Participants Receiving Concomitant Fluzone HD and CD388 Compared to Participants Who Receive Fluzone HD and Placebo | On Day 1 (pre-intervention baseline), Day 15 (±1 day), and Day 29/End of Trial (EOT) (±2 days)
  Evaluation of immune responses at 2- and 4-weeks post intervention measured by hemagglutinin inhibition (HAI) titers (geometric mean titers [GMTs] and seroconversion rates) against the influenza strains contained in the vaccine among participants receiving concomitant Fluzone HD influenza vaccine and CD388 compared to participants who receive Fluzone HD and placebo for CD388.

SECONDARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) in Participants Receiving Concomitant Fluzone HD and CD388 Compared to Participants Who Receive Fluzone HD and Placebo | From Day 1 through Day 29/EOT after concomitant intervention administration
  Safety and tolerability of CD388 will be evaluated by assessing the number of participants with incidences of TEAEs following the concomitant administration of either Fluzone HD influenza vaccine plus CD388 study drug or Fluzone HD plus placebo. TEAEs include but are not limited to adverse events (AEs), serious adverse events (SAEs), local adverse reactions (injection site reactions [ISRs]), systemic adverse reactions (myalgia, malaise, headache, and fever), and any potentially clinically significant changes from baseline seen in vital signs and clinical laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Davarpanah, MD, JD, Study Director — Cidara Therapeutics Inc.
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group (CCTMG) managed by Parexel, Glendale, California
  - Parexel International - EPCU Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No